CLINICAL TRIAL: NCT00887887
Title: The Association Between Gene Polymorphisms in the Innate Immune Response and the Risk of Infectious Complications and Liver Failure After Partial Hepatic Resection
Brief Title: The Association Between Gene Polymorphisms and Infectious Complications After Liver Surgery
Status: Completed | Type: Observational
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 08-4-022
Record Dates: First submitted 2009-04-23; First posted 2009-04-24 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Liver Disease
Keywords: liver surgery; gene polymorphisms; innate immune response; infectious complications; post-resectional liver failure; mortality
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, fresh frozen liver tissue
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- liver surgery: patients with benign or malignant hepatobiliary disease requiring partial hepatic resection

SUMMARY:
The purpose of the study is to test whether the presence of polymorphisms in genes encoding substances of the innate immune response in patients undergoing partial hepatic resection because of benign or malignant hepatobiliary disease is related to a higher incidence of infectious complications, post-resectional liver failure or mortality.

DETAILED DESCRIPTION:
Partial hepatic resection is a feasible and relatively safe procedure for selected patients with benign or malignant hepatobiliary disease. Liver failure after partial hepatic resection, so-called post-resectional liver failure (PLF), is a dreaded complication with high mortality rates. Patients suffering from PLF experience significantly more clinically significant infections (CSI) when compared with patients without PLF. The liver plays an important role in the body's innate immune defense. Recently, polymorphisms in genes encoding key molecules in the innate immune response (e.g. nuclear factor kappa-B) have shown to be associated with a greater risk of CSI. The presence of these polymorphisms combined with partial hepatic resection might render patients susceptible to the development of CSI, PLF and early mortality after liver resection.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* benign or malignant liver disease requiring partial hepatic resection

Exclusion Criteria:

* inability to give informed consent
* liver disease judged irresectable after intra-operative evaluation
* use of immunosuppressive drugs
* resection < 1 segment
* unable to comply with follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with benign or malignant liver disease requiring partial hepatic resection at the Maastricht University Medical Centre
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
clinically significant infectious complications (i.e. wound infection, pneumonia, blood stream infection, gastro-intestinal infection, intra-abdominal infection, urinary tract infection and miscellaneous) | 90 days after liver surgery

SECONDARY OUTCOMES:
post-resectional liver failure | 90 days after liver surgery
mortality | 90 days after liver surgery

CONTACTS AND LOCATIONS:
Overall Officials: Steven WM Olde Damink, MD, PhD, MSc, Principal Investigator — Maastricht University Medical Centre
Locations (1):
- Department of Surgery, Maastricht University Medical Centre, Maastricht, Netherlands